CLINICAL TRIAL: NCT03336684
Title: Evaluation of Rheumatoid Arthritis Disease Education Literature: The ERADEL Trial
Brief Title: Evaluation of Rheumatoid Arthritis Disease Education Literature
Acronym: ERADEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Atta Abbas Naqvi, Research Assistant, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PACT2
Record Dates: First submitted 2017-10-31; First posted 2017-11-08 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Patient education; Rheumatoid arthritis; Knowledge; Attitudes; Practice
MeSH Terms: conditions — Arthritis, Rheumatoid; Behavior | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator will be blinded from randomization and recruitment process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Education Group (Experimental): Patients will be provided with disease education literature
  Interventions: Behavioral: Patient education
- Normal Group (No Intervention): Patients will not be provided with disease education literature

INTERVENTIONS:
Behavioral: Patient education — Rheumatoid arthritis patients will be provided with disease education literature
  Arms: Patient Education Group

SUMMARY:
Rheumatoid arthritis is an inflammatory disease that results in joint inflammation, pain and swelling. It may progress to advance stages that render patients unable to carry out their daily activities. It also results in joints deformity and is a leading cause of disability globally.

Patient education plays an important role in the management of disease. Adequate patient knowledge and awareness about disease may help in incorporating the ailment in daily life. The purpose of this study is to evaluate the benefit of a disease education literature in Urdu language and with culturally relevant illustration for rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Out-patients with established diagnosis of rheumatoid arthritis over 3 months.
2. Participants who are willing to participate in the study.

Exclusion Criteria:

1. Patients with no rheumatoid arthritis.
2. Patients currently undergoing surgery or had previous history of surgery.
3. Patients who are not willing to participate.
4. In-patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Patient knowledge about rheumatoid arthritis | 3 months
  Measurement of patient's knowledge and awareness about rheumatoid arthritis using The 13-item Rheumatoid Arthritis Knowledge Assessment Scale (RAKAS-13) before and after the intervention.
  The RAKAS-13 is a psychometric tool consisting of 13 multiple choice questions related to rheumatoid arthritis disease knowledge. All questions have 1 point for "Right" answer and zero (0) points for "Wrong" answer.
  The scoring criteria are as follows:
  Excellent knowledge More than 75% correct answers = Above 11 points
  Adequate knowledge More than 50% or equal to 75% correct answers = 8 - 10 points
  Low knowledge More than 30% or equal to 50% correct answers = 5 - 7 points
  Poor knowledge Less than 30% correct answers = 4 points or less.

SECONDARY OUTCOMES:
Patient satisfaction | 3 months
  Patient satisfaction with be documented after the educational intervention using a patient satisfaction feedback form. It contains 10 questions related to general satisfaction from the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mehfooz Alam, MBBS, Principal Investigator — Liaqat National Hospital Karachi; Baqir S Naqvi, PhD, Study Director — Hamdard University
Locations (2):
- Pakistan (2):
  - Clifton Central Hospital, Karachi, Sindh
  - Liaqat National Hospital, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No